CLINICAL TRIAL: NCT02834065
Title: Cognitive Effects of Body Temperature During Hypothermic Circulatory Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Emory Healthcare (Other); University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH); Baylor Scott and White Health (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00064962; 1R01HL130443-01A1 (NIH)
Record Dates: First submitted 2016-07-06; First posted 2016-07-15 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cognition Disorders
Keywords: Postoperative Cognitive Decline; Deep Hypothermic Circulatory Arrest; Cardiovascular Surgical Procedures; Functional Magnetic Resonance Imaging; Small Ubiquitin-Related Modifier Proteins
MeSH Terms: conditions — Cognition Disorders; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep Hypothermia (Active Comparator): Initiation of circulatory arrest using the cardiopulmonary bypass machine at temperature ≤20 degrees Celsius
  Interventions: Device: Cardiopulmonary bypass machine
- Low Hypothermia (Active Comparator): Initiation of circulatory arrest using the cardiopulmonary bypass machine at temperature 20.1 - 24.0 degrees Celsius
  Interventions: Device: Cardiopulmonary bypass machine
- Moderate Hypothermia (Active Comparator): Initiation of circulatory arrest using the cardiopulmonary bypass machine at temperature 24.1 - 28 degrees Celsius
  Interventions: Device: Cardiopulmonary bypass machine

INTERVENTIONS:
Device: Cardiopulmonary bypass machine — Routinely used cardiopulmonary bypass machine (standard of care) will be used to initiate circulatory arrest

SUMMARY:
In this study the investigator will randomize 273 subjects to deep (<20°C), low (20.1°C-24°C), or moderate (24.1°C-28°C) hypothermia during aortic arch surgery with circulatory arrest. The primary purpose of this study is to determine the effect of deep vs low vs moderate hypothermia on neurocognitive function, brain functional connectivity, and leukocyte SUMOylation patterns after surgical circulatory arrest in participants.

DETAILED DESCRIPTION:
Purpose of the Study: Determine the effect of deep vs low vs moderate hypothermia on neurocognitive function, brain functional connectivity, and leukocyte SUMOylation patterns after surgical circulatory arrest.

Hypothesis: Deep hypothermia is superior to moderate hypothermia in reducing postoperative cognitive decline and preserving brain functional connectivity and that low hypothermia is non-inferior to deep hypothermia.

Design and Procedures: 273 informed and consenting patients who are scheduled for elective proximal aortic reconstructive surgery (ascending aorta + aortic valve or root) with concomitant proximal hemi- or total arch replacement via median sternotomy will be randomized to deep (<20°C), low (20.1°C-24°C), or moderate (24.1°C-28°C) hypothermia during circulatory arrest. Cognitive testing using a standard battery will occur preoperatively (baseline), at 4 weeks, and at 1 year after surgery. Neuroimaging procedures before surgery, and at 4 weeks and 1 year after surgery will consist of high-resolution anatomic, resting-state fMRI (rs-fMRI) and magnetic resonance spectroscopy (MRS) sequences. To characterize leukocyte activation, whole blood will be drawn at 5 time points: at baseline (prior to surgery), before circulatory arrest, 10 minutes after reperfusion, 10 minutes after CPB, and 4 hours after CPB.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective proximal aortic reconstructive surgery (ascending aorta + aortic valve or root) with concomitant proximal hemi- or total arch replacement via median sternotomy

Exclusion Criteria:

* < 18 years of age
* History of symptomatic cerebrovascular disease, eg, prior stroke with residual deficit
* Alcoholism (> 2 drinks/day)
* Psychiatric illness (any clinical diagnoses requiring therapy)
* Drug abuse (any illicit drug use in the past 3 months)
* Hepatic insufficiency (liver function tests > 1.5 times the upper limit of normal)
* Severe pulmonary insufficiency (requiring home oxygen therapy)
* Renal failure (serum creatinine > 2.0 mg/dL)
* Claustrophobic fear
* Unable to read and thus unable to complete the cognitive testing
* Pregnant women
* Patients who score < 24 on a baseline Mini Mental State Examination (MMSE) or ≥ 27 on the baseline Center for Epidemiological Studies Depression (CES-D) scale
* Patients who have pre-existing unsafe implants for 3 Tesla magnetic resonance imaging (MRI).
* Patients who have received chemotherapy in the last 12 months.
* Patients with COVID-19 diagnosis within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Change in short-term cognition as measured by continuous cognitive score | From baseline to 4 weeks post-operatively
  To characterize cognitive function over time while minimizing potential redundancy in the cognitive measures, a factor analysis will be performed on the cognitive test scores from baseline. A continuous change score will be calculated by subtracting the baseline cognitive index (the mean of the domain scores from factor analysis) from the follow-up cognitive index at 4 weeks.

SECONDARY OUTCOMES:
Change in SUMO 2/3 levels | Pre-incision, before circulatory arrest, 10 minutes after reperfusion, 10 minutes after cardiopulmonary bypass, 4 hrs after cardiopulmonary bypass
Change in long-term cognition as measured by continuous cognitive score | From baseline to 1 year post-operatively
  To characterize cognitive function over time while minimizing potential redundancy in the cognitive measures, a factor analysis will be performed on the cognitive test scores from baseline. A continuous change score will be calculated by subtracting the baseline cognitive index (the mean of the domain scores from factor analysis) from the follow-up cognitive index at 1 year.
Incidence of delirium | Up to post-operative day 3
  Confusion Assessment Method (CAM)
Change in neurological function as measured by NIHSS | Assessed at baseline, post-op day 4, 4 weeks
Change in neuronal metabolism | From baseline to 4 weeks
  Magnetic resonance spectra (metabolic peaks) of myoinositol, creatine, choline and N-acetyl aspartate
Change in resting-state functional connectivity | From baseline to 4 weeks post-operatively
  For the rs-fMRI data, the analyses of primary interest will be the spontaneous, low-frequency fluctuations in the blood oxygen level dependent (BOLD) data of the Default Mode, Salience, and Executive Control Networks.
Change in Duke Activity Status Index score | From baseline to 4 weeks postoperatively
Change in depression score | From baseline to 4 weeks postoperatively
  Measured by the Center for Epidemiological Studies Depression Scale (CES-D).
Change in anxiety score | From baseline to 4 weeks postoperatively
  Measured by State Trait Anxiety Inventory (STA-I).
Change in SF-36 score | From baseline to 1 year postoperatively
Change in employment status | From baseline to 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Mathew, MD, MHSc, MBA, Principal Investigator — Duke Health
Locations (4):
- United States (4):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Duke University Health System, Durham, North Carolina
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes GC, Chen EP, Browndyke JN, Szeto WY, DiMaio JM, Brinkman WT, Gaca JG, Blumenthal JA, Karhausen JA, Bisanar T, James ML, Yanez D, Li YJ, Mathew JP. Cognitive Effects of Body Temperature During Hypothermic Circulatory Arrest Trial (GOT ICE): A Randomized Clinical Trial Comparing Outcomes After Aortic Arch Surgery. Circulation. 2024 Feb 27;149(9):658-668. doi: 10.1161/CIRCULATIONAHA.123.067022. Epub 2023 Dec 12. PMID 38084590